CLINICAL TRIAL: NCT07000409
Title: The Effectiveness of Ultra-Sound Guided Erector Spinae Block With Betamethasone for Management of Truncal Chronic Post Herpetic Neuralgia, a Prospective Randomized Controlled Study.
Brief Title: The Effectiveness of Ultra-Sound Guided Erector Spinae Block With Betamethasone for Management of Truncal Chronic Post Herpetic Neuralgia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Refaat Eid, Assistant lecturer of Anesthesia, surgical ICU and pain management, Faculty of medicine, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-261-2024
Record Dates: First submitted 2025-05-24; First posted 2025-06-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Postherpetic Neuralgia; Chronic Pain; Ultrasound Guidance; Erector Spinae Plane Block; Betamethasone
MeSH Terms: conditions — Neuralgia, Postherpetic; Chronic Pain | interventions — Amitriptyline; Parapsychology; Dental Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Med group (Active Comparator): Patients will receive the standard medical regimen alone.
  Interventions: Other: Medical management regimen
- Erector spinae plane block group (Experimental): Patients will receive erector spinae plane (ESP) block with betamethasone with standard medical regimen.
  Interventions: Other: Erector spinae plane (ESP) block

INTERVENTIONS:
Other: Medical management regimen — Patients will receive the standard medical regimen alone.
  Other Names: Paracetamol +-Gabapentin + Amitriptyline
  Arms: Med group
Other: Erector spinae plane (ESP) block — Patients will receive erector spinae plane (ESP) block with betamethasone with standard medical regimen.
  Arms: Erector spinae plane block group

SUMMARY:
To investigate the effectiveness of ultra-Sound guided Erector spinae block (ESB) with Betamethasone as an adjuvant to standard medical protocol in the management of truncal chronic post herpetic neuralgia.

DETAILED DESCRIPTION:
Postherpetic neuralgia (PHN) is a syndrome described as zoster-associated pain persisting for more than 3 months after resolution of an initial herpes zoster (HZ) rash ("shingles").[This condition is considered to be the most prevalent and challenging complication associated with HZ infection. According to reports, around 75% of senior patients who contract HZ are likely to experience it. The incidence of it was observed to be 38.1%, 27.0%, and 19.0% at 1 month, 3 months, and 6 months, respectively, following the onset of zoster. Half of the patients who are more than 50 years have the risk of developing PHN. It is noteworthy that the incidence of PHN seems to be on the rise.

Erector spinae plane (ESP) block is one of the newer interfascial techniques where the drug is injected below the erector spinae muscle to spread towards the costotransverse foramina and origin of dorsal and ventral rami where it is supposed to work at the origin of spinal nerves, based on cadaveric and contrast studies. Cadaveric studies have also showed that a block at T5 level is sufficient to have unilateral multi-dermatomal sensory block ranging from T1 to L3. Thus, this block serves the purpose of a paravertebral block without the risk of pleural injury.

Betamethasone is a long-acting corticosteroid with immunosuppressive and anti-inflammatory properties. It can be used topically to manage inflammatory skin conditions such as eczema, and parenterally to manage several disease states including autoimmune disorders. Betamethasone has potent glucocorticoid activity and negligible mineralocorticoid activity. The beneficial effects of injecting steroids could be because of sympathetic blockage, thereby inhibiting vasoconstriction and due to anaesthetization of the dorsal root ganglion and posterior spinal nerve.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18 and 75.
* Patients with American Society of Anesthesiologists (ASA) II and III status.
* Patients diagnosed with truncal chronic post herpetic neuralgia( neuropathic pain persistent for more than 3 months from the onset of rash appearance )

Exclusion Criteria:

* Patients unable to comprehend the informed consent.
* Patients on long term opioid regimens.
* Patients with impairment in hepatic (Alanine aminotransferase (ALT) >50 U/L, and/or Aspartate aminotransferase (AST): >45 U/L) or renal functions( creatinine level ≥1.5 mg/dL)
* Patients on anti-coagulation regimens.
* Patients with coagulation abnormalities (i.e. international normalized ratio (INR) ≥1.5 and/or platelets ≤50000)
* Local infection in the site of the block.
* Patients with body mass index (BMI) > 35.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain degree | 8 weeks after the first clinic visit.
  The degree of pain will be obtained and recorded on a numeric rating scale (NRS) with 0=no pain, and 10=Maximum pain intensity. Pain NRS score will be assessed at 2,4,6,8 weeks after the first clinic visit.

SECONDARY OUTCOMES:
Incidence of side effects | 8 weeks after the first clinic visit.
  Incidence of side effects for medications regimen (excessive sleepiness, nausea, vomiting allergic reaction, diarrhea, blurred vision, disorientation).
Incidence of side effects | 8 weeks after the first clinic visit.
  Incidence of side effects for ESP block (local hematoma, limb numbness or weakness, dizziness, pneumothorax, hypotension, infection, allergic reaction).
Tramadol consumption in both groups. | 8 weeks after the first clinic visit.
  Total consumption of tramadol in both groups will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.